CLINICAL TRIAL: NCT02171988
Title: Comparison of Effect of Propranolol, Bisoprolol, Pyridosgitmine in Postural Orthostatic Tachycardia Syndrome (POTS) and Prognosis After Medical Treatment
Brief Title: Effect of Medical Treatment and Prognosis of Postural Orthostatic Tachycardia Syndrome (POTS)
Acronym: POTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, MD, PhD, professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1401091550
Record Dates: First submitted 2014-06-19; First posted 2014-06-24 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: Postural Orthostatic Tachycardia Syndrome; propranolol; bisoprolol; pyridostigmine
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Propranolol; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Propranolol (Active Comparator): Start propranolol 10mg bid, and then dose up to 20mg bid after one month if tolerable
  Interventions: Drug: Propranolol
- Bisoprolol (Active Comparator): Start bisoprolol 2.5mg qd P.O, and then dose up to 5mg qd. if tolerable
  Interventions: Drug: Bisoprolol
- Propranolol+pyridostigmine (Active Comparator): Start propranolol+pyridostigmine 10mg bid +30mg bid, and then dose up to 20mg bid+30mg bid. if tolerable.
  Interventions: Drug: Propranolol+pyridostigmine
- Bisoprolol+pyridostgmine (Active Comparator): start bisoprolol+pyridostgmine 2.5mg qd+30mg bid, and then, dose up to 5mg qd+30mg bid. if tolerable
  Interventions: Drug: Bisoprolol+pyridostgmine

INTERVENTIONS:
Drug: Propranolol — Start propranolol 10mg bid, and then dose up to 20mg bid after one month if tolerable
  Arms: Propranolol
Drug: Bisoprolol — Start bisoprolol 2.5mg qd P.O, and then dose up to 5mg qd. if tolerable
  Arms: Bisoprolol
Drug: Propranolol+pyridostigmine — Start propranolol+pyridostigmine 10mg bid +30mg bid, and then dose up to 20mg bid+30mg bid. if tolerable.
  Arms: Propranolol+pyridostigmine
Drug: Bisoprolol+pyridostgmine — Start bisoprolol+pyridostgmine 2.5mg qd+30mg bid, and then, dose up to 5mg qd+30mg bid. if tolerable
  Arms: Bisoprolol+pyridostgmine

SUMMARY:
The purpose of the study is to investigate effect of medical treatment and prognosis of Postural Orthostatic Tachycardia Syndrome (POTS)

DETAILED DESCRIPTION:
Many patients who complained of dizziness are eventually diagnosed as POTS. However, the investigation of an appropriate medical treatment of POTS has not been enough yet. Also, the prognosis of the disease after treatment is not well known. It is known that propranolol attenuate the tachycardia and improve symptom burden in patients with POTS. However, the effect of other β-Blocker, bisoprolol compared with propranolol is not known well. In addition, acetylcholinesterase inhibition with pyridostigmine was a effective method of acutely decreasing the tachycardia in patients with POTS. However, difference among three medical treatments effect is not known and long-term studies are not done yet. Therefore, in this study investigator investigate effect of medical treatment (propranolol only, bisoprolol only, propranolol+pyridostigmine, bisoprolol+pyridostigmine) and prognosis of Postural Orthostatic Tachycardia Syndrome.

Longer-term studies are needed to assess this promising therapy.

ELIGIBILITY:
Inclusion Criteria:

* aged 15<=
* developed symptoms of orthostatic intolerance accompanied by a HR rise ≥30 min-1 within the first 10 minutes of standing, HR rise ≥ 120 in the absence of orthostatic hypotension (a fall in blood pressure [BP] >20/10 mm Hg).

Exclusion Criteria:

* poor drug compliance
* patients who cannot or do not want to write questionaires.
* patients who do not want draw blood

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The change of the subjective symptom survey result after 3-month medical treatment. | 3 month after medical treatment

SECONDARY OUTCOMES:
Normalization of orthostatic BP-HR test after 6-month medical treatment. | 6 month
The change of the subjective symptom after 6-month medical treatment. | 6 month
Change of quality of life score after treatment | 6 month
Change of depression score after treatment | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Kon Chu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Raj SR, Black BK, Biaggioni I, Harris PA, Robertson D. Acetylcholinesterase inhibition improves tachycardia in postural tachycardia syndrome. Circulation. 2005 May 31;111(21):2734-40. doi: 10.1161/CIRCULATIONAHA.104.497594. Epub 2005 May 23. PMID 15911704
- [Background] Raj SR, Black BK, Biaggioni I, Paranjape SY, Ramirez M, Dupont WD, Robertson D. Propranolol decreases tachycardia and improves symptoms in the postural tachycardia syndrome: less is more. Circulation. 2009 Sep 1;120(9):725-34. doi: 10.1161/CIRCULATIONAHA.108.846501. Epub 2009 Aug 17. PMID 19687359
- [Background] Fu Q, Vangundy TB, Shibata S, Auchus RJ, Williams GH, Levine BD. Exercise training versus propranolol in the treatment of the postural orthostatic tachycardia syndrome. Hypertension. 2011 Aug;58(2):167-75. doi: 10.1161/HYPERTENSIONAHA.111.172262. Epub 2011 Jun 20. PMID 21690484
- [Background] Kimpinski K, Figueroa JJ, Singer W, Sletten DM, Iodice V, Sandroni P, Fischer PR, Opfer-Gehrking TL, Gehrking JA, Low PA. A prospective, 1-year follow-up study of postural tachycardia syndrome. Mayo Clin Proc. 2012 Aug;87(8):746-52. doi: 10.1016/j.mayocp.2012.02.020. Epub 2012 Jul 15. PMID 22795533
- [Background] Sousa A, Lebreiro A, Freitas J, Maciel MJ. Long-term follow-up of patients with postural tachycardia syndrome. Clin Auton Res. 2012 Jun;22(3):151-3. doi: 10.1007/s10286-011-0155-1. Epub 2011 Dec 22. PMID 22190289
- [Background] Winker R, Barth A, Bidmon D, Ponocny I, Weber M, Mayr O, Robertson D, Diedrich A, Maier R, Pilger A, Haber P, Rudiger HW. Endurance exercise training in orthostatic intolerance: a randomized, controlled trial. Hypertension. 2005 Mar;45(3):391-8. doi: 10.1161/01.HYP.0000156540.25707.af. Epub 2005 Feb 7. PMID 15699447
- [Background] Arnold AC, Okamoto LE, Diedrich A, Paranjape SY, Raj SR, Biaggioni I, Gamboa A. Low-dose propranolol and exercise capacity in postural tachycardia syndrome: a randomized study. Neurology. 2013 May 21;80(21):1927-33. doi: 10.1212/WNL.0b013e318293e310. Epub 2013 Apr 24. PMID 23616163
- [Background] Benarroch EE. Postural tachycardia syndrome: a heterogeneous and multifactorial disorder. Mayo Clin Proc. 2012 Dec;87(12):1214-25. doi: 10.1016/j.mayocp.2012.08.013. Epub 2012 Nov 1. PMID 23122672
- [Background] Mathias CJ, Low DA, Iodice V, Owens AP, Kirbis M, Grahame R. Postural tachycardia syndrome--current experience and concepts. Nat Rev Neurol. 2011 Dec 6;8(1):22-34. doi: 10.1038/nrneurol.2011.187. PMID 22143364
- [Derived] Moon J, Kim DY, Lee WJ, Lee HS, Lim JA, Kim TJ, Jun JS, Park B, Byun JI, Sunwoo JS, Lee ST, Jung KH, Park KI, Jung KY, Kim M, Lee SK, Chu K. Efficacy of Propranolol, Bisoprolol, and Pyridostigmine for Postural Tachycardia Syndrome: a Randomized Clinical Trial. Neurotherapeutics. 2018 Jul;15(3):785-795. doi: 10.1007/s13311-018-0612-9. PMID 29500811